CLINICAL TRIAL: NCT03190616
Title: A Single Arm, Open Label, Multicenter Exploratory Study of Apatinib in Patients With Metastatic Colorectal Cancer (CRC) Who Have Progressed After Standard Second Line Therapy
Brief Title: Apatinib in Refractory Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry); Beijing gene plus technology co., LTD (Unknown)
Responsible Party: Principal Investigator, Gu Yanhong, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEEP-G 01
Record Dates: First submitted 2017-03-01; First posted 2017-06-19 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- drug,apatinib (Experimental): apatinib 500mg/qd, 28d/cycle
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: apatinib — apatinib 500mg/qd, 28d/cycle
  Other Names: YN968D1

SUMMARY:
Limited agents have been approved after standard first and second line treatment. Regorafenib and Trifluridine/Tipiracil (TAS-102) are still not approved in China.Apatinib has shown significant efficacy in refractory advanced gastric cancer regarding PFS and OS with controllable toxicity.This study is aimed to explore the efficacy,safety as well as predictive biomarker in advanced colorectal cancer failed to standard therapy in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.
* Subjects with metastatic colorectal cancer(CRC) (Stage IV).
* Subjects must have failed at least two lines of prior treatment, which must include a fluoropyrimidine, oxaliplatin and irinotecan.
* Subjects treated with oxaliplatin in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy.
* Subjects who have withdrawn from standard treatment due to unacceptable toxicity and precluding retreatment with the same agent prior to progression of disease will also be allowed.
* Prior treatment with bevacizumab and/or cetuximab will be allowed.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.is necessary.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Life expectancy of at least 3 months.
* Adequate bone marrow, liver and renal function as assessed by the laboratory required by protocol.
* assigned informed consent.

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Participants of other clinical trial within 4 weeks.
* Diseases which will impact the absorption of apatinib, eg. dysphagia, chronic diarrhea, bowl obstruction
* Hemorrhage events of ≥grade 3 within 4 weeks.
* known central nervous system metastasis.
* Uncontrolled hypertension. (Systolic blood pressure 140 mmHg or diastolic pressure 90 mmHg despite optimal medical management). Unstable angina,congestive heart failure,Myocardial infarction, Cardiac arrhythmias requiring anti-arrhythmic therapy.
* urine protein ≥++ and 24h urine protein more than 1.0g.
* Chronically green wound or bone fracture.
* Arterial or venous thrombotic or embolic events.
* Tumor invading important blood vessel with high risk of severe hemorrhage.
* Abnormal coagulation function.
* thromboemboli events within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival(PFS) | From assignment of the first subject to 3 months later after the last participant is recruited.The last participant will be recruited before Mar 30,2019
  PFS was defined as the time from assignment to disease progression radiological/clinical or death due to any cause, whichever occurs first. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation.

SECONDARY OUTCOMES:
Overall Survival (OS) | From assignment of the first subject until 40 death events observed, up to 2 years.
  OS is defined as the time from date of assignment to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Disease control rate (DCR) | From assignment of the first subject to 3 months later after the last participant is recruited.The last participant will be recruited before Mar 30,2019
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD)
Objective response rate(ORR) | From assignment of the first subject to 3 months later after the last participant is recruited.The last participant will be recruited before Mar 30,2019
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR)
Quality of life | From assignment of the first subject to 3 months later after the last participant is recruited.The last participant will be recruited before Mar 30,2019
  The general well-being of participants, outlining negative and positive features of life.
relationship between the tumor molecular burden & gene mutation and the drug efficacy. | From assignment of the first subject to 3 months later after the last participant is recruited.The last participant will be recruited before Mar 30,2019.
  The tumor molecular clones and gene mutations of 1021 tumor related genes will be detected by next-generation sequencing,which will be matched with the CT scanning .
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From assignment of the first subject to 3 months later after the last participant is recruited.The last participant will be recruited before Mar 30,2019.
  adverse events will be assessed according to CTCAE v4.0, including hematological and non-hematological adverse events. Non-hematological adverse events will be collected by patients reported outcomes questionaire. The adverse events of interest include hypertension,hand-foot syndrome,proteinuria,hoarseness,rash,etc.The dose reduction and drug discontinuance due to adverse events will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Gu, Dr., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (4):
- China (4):
  - the second hospital of Changzhou city, Changzhou, Jiangsu
  - Nanjing 81 Hospital, Nanjing, Jiangsu
  - the first affiliated hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Jiangnan University affiliated hospital, Wuxi, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Background] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952